CLINICAL TRIAL: NCT00519259
Title: Tolerability, Safety, and Pharmacokinetics of Repeated Sublingual Doses of Lobeline
Brief Title: Tolerability and Safety of 30, 45, and 60 mg of Sublingual Lobeline. - 1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-CPU-0009-1
Record Dates: First submitted 2006-06-29; First posted 2007-08-22 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2006-06

CONDITIONS: Methamphetamine Dependence
MeSH Terms: interventions — Lobeline

INTERVENTIONS:
Drug: Lobeline

SUMMARY:
The purpose of this study is to assess safety and pharmacokinetics of sublingual lobeline in healthy normal volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to provide written informed consent
* Must have a body mass index between 18 and 30
* Have no medical contraindications as determined by medical history, physical exam, ECG, hematology and blood chemistry profile, and urinalysis
* Must have a negative drug test at screening and admission
* If female of child bearing potential, must agree to use birth control

Exclusion Criteria:

* Please contact the site for more information

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12
Dates: Start 2006-02

PRIMARY OUTCOMES:
Tolerability

SECONDARY OUTCOMES:
Safety
Pharmacokinetic parameters
Cardiovascular responses
Psychological effects of lobeline

CONTACTS AND LOCATIONS:
Overall Officials: Reese Jones, M.D., Principal Investigator — Langley Porter Psychiatric Institute
Locations (1):
- Langley Porter Psychiatric Institute, San Francisco, California, United States